CLINICAL TRIAL: NCT02267837
Title: OrthoPulse™ and Its Effect on the Rate of Orthodontic Tooth Alignment: A Pilot Feasibility Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biolux Research Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TS1.5
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Results first posted 2015-09-11 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Malocclusion
Keywords: Alignment phase; Photobiomodulation; Orthodontic treatment; Malocclusion; OrthoPulse™
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OrthoPulse™ (Experimental): Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Interventions: Device: OrthoPulse™
- Control (No Intervention): Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment only, and no OrthoPulse™ treatments.

INTERVENTIONS:
Device: OrthoPulse™ — Patients carry out daily OrthoPulse™ treatments at home.
  Arms: OrthoPulse™

SUMMARY:
The aim of this study is to determine the effect of OrthoPulse™, an intra-oral LED (Light Emitting Diode) photobiomodulation device, on the rate of anterior orthodontic alignment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of permanent dentition
* Eligible and scheduled for full mouth fixed orthodontic treatment
* Class I or Class II malocclusion (no more than ½ cusp in Class II)
* Non-extraction in all quadrants
* Non-smoker
* Good oral hygiene as determined by the investigator
* No adjunct treatment such as extra- or intra-oral appliances

Exclusion Criteria:

* Pregnant females
* Patient is currently enrolled in another clinical study
* Non-steroidal Anti-Inflammatory drug (NSAID) use during study (Acetominophen acceptable)
* Periodontally involved teeth
* Use of bisphosphonates
* Unerupted or partially erupted maxillary teeth
* Teeth blocked out of alignment and unable to engage initial arch wire
* Spaces present in the maxillary arch

Ages: 11 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Shaughnessy, DDS, Principal Investigator — Shaughnessy Orthodontics
Locations (1):
- Shaughnessy Orthodontics, Suwanee, Georgia, United States

REFERENCES:
- [Background] Nimeri G, Kau CH, Corona R, Shelly J. The effect of photobiomodulation on root resorption during orthodontic treatment. Clin Cosmet Investig Dent. 2014 Jan 15;6:1-8. doi: 10.2147/CCIDE.S49489. eCollection 2014. PMID 24470774
- [Background] Ekizer A, Uysal T, Guray E, Akkus D. Effect of LED-mediated-photobiomodulation therapy on orthodontic tooth movement and root resorption in rats. Lasers Med Sci. 2015 Feb;30(2):779-85. doi: 10.1007/s10103-013-1405-3. Epub 2013 Aug 29. PMID 23990217
- [Background] El-Bialy T, Alhadlaq A, Felemban N, Yeung J, Ebrahim A, Hassan AH. The effect of light-emitting diode and laser on mandibular growth in rats. Angle Orthod. 2015 Mar;85(2):233-8. doi: 10.2319/030914-170.1. Epub 2014 Jul 14. PMID 25017014
- [Background] Uysal T, Ekizer A, Akcay H, Etoz O, Guray E. Resonance frequency analysis of orthodontic miniscrews subjected to light-emitting diode photobiomodulation therapy. Eur J Orthod. 2012 Feb;34(1):44-51. doi: 10.1093/ejo/cjq166. Epub 2010 Dec 27. PMID 21187526
- [Background] Ekizer A, Uysal T, Guray E, Yuksel Y. Light-emitting diode photobiomodulation: effect on bone formation in orthopedically expanded suture in rats--early bone changes. Lasers Med Sci. 2013 Sep;28(5):1263-70. doi: 10.1007/s10103-012-1214-0. Epub 2012 Nov 9. PMID 23139069
- [Background] Kau CH, Kantarci A, Shaughnessy T, Vachiramon A, Santiwong P, de la Fuente A, Skrenes D, Ma D, Brawn P. Photobiomodulation accelerates orthodontic alignment in the early phase of treatment. Prog Orthod. 2013 Sep 19;14:30. doi: 10.1186/2196-1042-14-30. PMID 24326198
- [Background] Dias FJ, Issa JP, Vicentini FT, Fonseca MJ, Leao JC, Siessere S, Regalo SC, Iyomasa MM. Effects of low-level laser therapy on the oxidative metabolism and matrix proteins in the rat masseter muscle. Photomed Laser Surg. 2011 Oct;29(10):677-84. doi: 10.1089/pho.2010.2879. Epub 2011 Jul 11. PMID 21745137
- [Background] Silveira PC, Silva LA, Fraga DB, Freitas TP, Streck EL, Pinho R. Evaluation of mitochondrial respiratory chain activity in muscle healing by low-level laser therapy. J Photochem Photobiol B. 2009 May 4;95(2):89-92. doi: 10.1016/j.jphotobiol.2009.01.004. Epub 2009 Jan 21. PMID 19232497
- [Background] Cruz DR, Kohara EK, Ribeiro MS, Wetter NU. Effects of low-intensity laser therapy on the orthodontic movement velocity of human teeth: a preliminary study. Lasers Surg Med. 2004;35(2):117-20. doi: 10.1002/lsm.20076. PMID 15334614
- [Background] Esper MA, Nicolau RA, Arisawa EA. The effect of two phototherapy protocols on pain control in orthodontic procedure--a preliminary clinical study. Lasers Med Sci. 2011 Sep;26(5):657-63. doi: 10.1007/s10103-011-0938-6. Epub 2011 May 31. PMID 21626017
- [Background] Youssef M, Ashkar S, Hamade E, Gutknecht N, Lampert F, Mir M. The effect of low-level laser therapy during orthodontic movement: a preliminary study. Lasers Med Sci. 2008 Jan;23(1):27-33. doi: 10.1007/s10103-007-0449-7. Epub 2007 Mar 15. PMID 17361391
- [Background] Sousa MV, Scanavini MA, Sannomiya EK, Velasco LG, Angelieri F. Influence of low-level laser on the speed of orthodontic movement. Photomed Laser Surg. 2011 Mar;29(3):191-6. doi: 10.1089/pho.2009.2652. Epub 2011 Jan 23. PMID 21254890
- [Background] Heravi F, Moradi A, Ahrari F. The effect of low level laser therapy on the rate of tooth movement and pain perception during canine retraction. Oral Health Dent Manag. 2014 Jun;13(2):183-8. PMID 24984620
- [Background] Whelan HT, Smits RL Jr, Buchman EV, Whelan NT, Turner SG, Margolis DA, Cevenini V, Stinson H, Ignatius R, Martin T, Cwiklinski J, Philippi AF, Graf WR, Hodgson B, Gould L, Kane M, Chen G, Caviness J. Effect of NASA light-emitting diode irradiation on wound healing. J Clin Laser Med Surg. 2001 Dec;19(6):305-14. doi: 10.1089/104454701753342758. PMID 11776448
- [Background] Weber JB, Pinheiro AL, de Oliveira MG, Oliveira FA, Ramalho LM. Laser therapy improves healing of bone defects submitted to autologous bone graft. Photomed Laser Surg. 2006 Feb;24(1):38-44. doi: 10.1089/pho.2006.24.38. PMID 16503787
- [Background] Saito S, Shimizu N. Stimulatory effects of low-power laser irradiation on bone regeneration in midpalatal suture during expansion in the rat. Am J Orthod Dentofacial Orthop. 1997 May;111(5):525-32. doi: 10.1016/s0889-5406(97)70152-5. PMID 9155812
- [Background] Masha RT, Houreld NN, Abrahamse H. Low-intensity laser irradiation at 660 nm stimulates transcription of genes involved in the electron transport chain. Photomed Laser Surg. 2013 Feb;31(2):47-53. doi: 10.1089/pho.2012.3369. Epub 2012 Dec 16. PMID 23240874
- [Background] Oron U, Ilic S, De Taboada L, Streeter J. Ga-As (808 nm) laser irradiation enhances ATP production in human neuronal cells in culture. Photomed Laser Surg. 2007 Jun;25(3):180-2. doi: 10.1089/pho.2007.2064. PMID 17603858
- [Background] Sun X, Zhu X, Xu C, Ye N, Zhu H. [Effects of low energy laser on tooth movement and remodeling of alveolar bone in rabbits]. Hua Xi Kou Qiang Yi Xue Za Zhi. 2001 Oct;19(5):290-3. Chinese. PMID 12539482
- [Derived] Shaughnessy T, Kantarci A, Kau CH, Skrenes D, Skrenes S, Ma D. Intraoral photobiomodulation-induced orthodontic tooth alignment: a preliminary study. BMC Oral Health. 2016 Jan 13;16:3. doi: 10.1186/s12903-015-0159-7. PMID 26762247

RESULTS

PARTICIPANT FLOW:
Groups:
- OrthoPulse™: Subjects assigned to this group receive fixed orthodontic appliance treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Full mouth fixed orthodontic appliance treatment: Patients are treated for full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
  OrthoPulse™: Patients carry out daily OrthoPulse™ treatments at home.
- No OrthoPulse™: Subjects assigned to this group receive fixed orthodontic appliance treatment only, and no OrthoPulse™ treatments.
  Full mouth fixed orthodontic appliance treatment: Patients are treated for full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
Period: Overall Study
Arm/Group | OrthoPulse™ | No OrthoPulse™
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OrthoPulse™: Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI), in conjunction with receiving daily OrthoPulse™ treatments. Treatment and follow-up appointments per the traditional practices of the PI and dental office.
  OrthoPulse™: Patients carry out daily OrthoPulse™ treatments at home.
- Control: Subjects assigned to this group receive only full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI), and no OrthoPulse™ treatments. Treatment and follow-up appointments per the traditional practices of the PI and dental office.
- Total: Total of all reporting groups
Arm/Group | OrthoPulse™ | Control | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 14.0 (1.7) | 15.0 (4.8) | 14.5 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Rate of Orthodontic Anterior Alignment in Millimetres Per Week (mm/wk) by Means of Little's Irregularity Index (LII) for OrthoPulse™ and Non-OrthoPulse™ Treated Patients.
Time Frame: Participants followed for the time it takes to complete orthodontic anterior alignment, an expected average of 30-120 days from the start of orthodontic treatment, depending on the severity of the case.
Measure: Mean (Standard Deviation); unit: millimeters per week (mm/wk)
Units Other Than Participants: arches
Groups:
- OrthoPulse™: Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment in conjunction with receiving daily OrthoPulse™ treatments.
  Full mouth fixed orthodontic appliance treatment: Patients are treated for full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
  OrthoPulse™: Patients carry out daily OrthoPulse™ treatments at home.
- No OrthoPulse™: Subjects assigned to this group receive full mouth fixed orthodontic appliance treatment only, and no OrthoPulse™ treatments.
  Full mouth fixed orthodontic appliance treatment: Patients are treated for full mouth fixed orthodontic appliance treatment by the qualified Principal Investigator (PI). Treatment and follow-up appointments per the traditional practices of the PI and dental office.
Arm/Group | OrthoPulse™ | No OrthoPulse™
Number analyzed (Participants) | 11 | 9
Number analyzed (arches) | 18 | 13
millimeters per week (mm/wk) | 1.27 (0.53) | 0.43 (0.20)

ADVERSE EVENTS:
Arm/Group | OrthoPulse™ | No OrthoPulse™
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No